CLINICAL TRIAL: NCT00595218
Title: How Can Radiation Oncologists Better Serve Their Patients? A Randomized Study to Determine Whether Radiation Oncologists Can Improve Patient Satisfaction by Attempting to Meet Their Patients' Preferences
Brief Title: Patient Preference Survey for Radiation Oncologists
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Dwight Heron, PI Mentor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: PittRadOnc; ASTRO grant
Record Dates: First submitted 2008-01-04; First posted 2008-01-16 (Estimated); Last update posted 2017-07-25 (Actual); Status verified 2017-07

CONDITIONS: Breast Cancer; Prostate Cancer; Lung Cancer
Keywords: Patient Preferences; Patient Satisfaction; Patient-Doctor Relationship
MeSH Terms: conditions — Breast Neoplasms; Prostatic Neoplasms; Lung Neoplasms; Patient Preference; Patient Satisfaction

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- 1 (No Intervention): Patients whose radiation oncologist are blinded to their patient preference survey results
- 2 (Active Comparator): Patients whose radiation oncologist are not blinded to their patient preference survey results
  Interventions: Behavioral: Physician behavior related to Patient Preference Survey; Other: Patient Preference Results

INTERVENTIONS:
Behavioral: Physician behavior related to Patient Preference Survey — Access to initial Patient preference survey results
  Arms: 2
Other: Patient Preference Results — Knowledge of Patient Preference Results
  Arms: 2

SUMMARY:
Limited data exists for the cancer patients' preferences on their patient-doctor interaction with their radiation oncologist. These physicians have the opportunity to develop intimate relationships with their patients since these patients typically require daily radiation treatments anywhere from one to seven weeks. Thus, by having a greater understanding of the individual patient preferences, the radiation oncologists will be able to better serve their patients leading to improved patient satisfaction with their physician and healthier outlook on life. This is the premise and the hypothesis of this study.

DETAILED DESCRIPTION:
An instrument, a questionnaire, previously developed by our group (IRB# 0512075) will be used to determine these cancer patient/subjects' preferences for the following six categories (see Appendix 1)

1. How should the radiation oncologist address them (by their first name or Mr/Mrs)?
2. Should the radiation oncologists wear a white coat?
3. Should the radiation oncologist discuss their prognosis and survival with them?
4. Should the radiation oncologist have physical contact with their patient (hold hand or hug the patient.)?
5. Should the radiation oncologist inquire about their religious beliefs to help cope with their cancer?
6. Should the radiation oncologist use basic, lay language or more technical terminology when describing the radiation treatment?

This research study will consist of a randomized study of breast, prostate, and lung cancer patients/subjects receiving radiation therapy at the University of Pittsburgh Cancer Institute and UPMC Cancer Centers who will complete this questionnaire. Radiation therapy can be either for definitive or palliative therapy. This creates six distinct cohorts in the study (definitive breast, prostate, and lung cancer, palliative breast, prostate, and lung cancer) that provide an adequate representation of the cancer patient/subject cohorts that receive radiation therapy.

Patients/subjects will answer this questionnaire at the time of the initial consultation with the radiation oncologist (before meeting the radiation oncologist), once midway during radiation therapy, and at the completion of the radiation treatment. At completion, there will be additional questions used from a modified version of an established validated instrument currently being used at the University of Pittsburgh Cancer Institute to assess patient/subject satisfaction. (Appendix 2). Participants will rate the importance of each item on a 5-point scale: strongly disagree, disagree, neither agree nor disagree, agree, or strongly agree. They will also use a parallel ranking from 0-100 on each item to more finely assess the satisfaction differences for the survey in Appendix 2 only.

After subjects answer the questionnaire at time of initial consultation, the subject will then be randomized to either an experimental or control group. In the experimental group, the radiation oncologist participants will read their patient's responses to this questionnaire prior to their initial consultation and try to adapt to the subject's (patient's) preferences. In the control group, the radiation oncologist participant will be blinded to the results of their patient's questionnaire. At the end of treatment, the radiation oncologists who viewed their patient preferences will have to answer the following question according to the 5 point scale system: "Did knowledge of your patient's preferences influence your behavior?" The radiation oncologist participant will not have access to the patient satisfaction survey.

The duration of study per patient participant will the duration of the radiation treatment which has an average length of 4 weeks. A subject accrual of 500 patient participants and 30 radiation oncologist participants is expected at the University of Pittsburgh Cancer Institute and UPMC Cancer Centers, consisting of 19 Radiation Oncology centers across Western Pennsylvania. The expected duration of the entire study is 1 year. The data will be collected through these instruments to generate a database collected in our database management system. The data will be coded and maintained by the clinical study coordinator.

ELIGIBILITY:
Inclusion Criteria:Any Patient/subject (adult male or female) with prostate or breast or lung cancer (Primary or Metastatic) who is scheduled to receive radiation therapy at one of the UPMC Cancer Centers

* Patient/subject must receive radiation treatment in addition to consultation with the Radiation Oncologist
* Patient/subject must meet with radiation oncologist at least one day per week while receiving radiation therapy.
* Any attending radiation oncologist whose patient is enrolled in this study

Exclusion Criteria:

* Patient/subject under age 18 If subject previously underwent this study, even if the previous study was for a different diagnosis. Subjects can only undergo this study once.

Patients/subjects who do not have the functional and mental capacity to independently answer the questionnaire.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2006-04; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Did knowledge of patient preference improve patient satisfaction | Length of radiation treatment

SECONDARY OUTCOMES:
Patient preferences regarding their radiation oncologists | Length of radiation treatment course

CONTACTS AND LOCATIONS:
Overall Officials: Ajay Bhatnagar, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- UPMC Cancer Centers, Pittsburgh, Pennsylvania, United States